CLINICAL TRIAL: NCT02781298
Title: Acceptability, Tolerance, Satiety and Prebiotic Effect of a New Infant Cereal in Infant Between 5 and 8 Months of Age, at the Beginning of Complementary Feeding
Brief Title: Acceptability, Tolerance, Satiety and Prebiotic Effect of a New Infant Cereal
Acronym: ACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hero Institute for Infant Nutrition (Industry)
Collaborators: Universidad de Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other); Quantum Experimental (Unknown)
Responsible Party: Principal Investigator, Luis Manuel Sanchez Siles, Director Innovation Infant Nutrition, Hero Institute for Infant Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT09-14
Record Dates: First submitted 2016-05-09; First posted 2016-05-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Infant Nutrition Sciences

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Infant Cereal (Experimental): amount ingested according to pediatricians recommendations
  Interventions: Dietary Supplement: New Infant Cereal; Dietary Supplement: Multicereals Infant Cereal
- Multicereals Infant Cereal (Active Comparator): amount ingested according to pediatricians recommendations
  Interventions: Dietary Supplement: New Infant Cereal; Dietary Supplement: Multicereals Infant Cereal

INTERVENTIONS:
Dietary Supplement: New Infant Cereal — The infants will start the complementary feeding with the infants cereals of this study, the amount of cereal ingested will be free according to pediatricians recommendations.
Dietary Supplement: Multicereals Infant Cereal — The infants will start the complementary feeding with the infants cereals of this study, the amount of cereal ingested will be free according to pediatricians recommendations.

SUMMARY:
This study evaluates a new infant cereals on acceptability, tolerance, satiety and prebiotic effect in infants.

DETAILED DESCRIPTION:
This is a controlled, randomized, prospective, crossover, triple-blind study to evaluate of a new infant cereal with a portion of whole grain flour on sensorial acceptability, gastrointestinal tolerance, satiety and prebiotic effect in healthy infants fron 5 to 8 months of age at the beginning of complementary feeding.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infant
* Birth weight 2500-4200 g
* Tolerance to cow's milk
* Tolerance to lactose
* No Breastfeeding at least 4 months of age
* No use antibiotic at least 2 weeks before recruitments

Exclusion Criteria:

* Intolerance to gluten (celiac disease)
* Congenital abnormalities
* Acute diseases
* Chronic situation that affect to food intake or metabolism
* Breastfeeding infant
* Any food allergy
* Participation in other study

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Hedonic scale- Sensorial Evaluation | Day 24, day 73
  Sensorial acceptability -Differences between groups measured by Hedonic scales (4-points for children and 7-points for adults)

SECONDARY OUTCOMES:
Weight | Day 1 (Baseline), Day 45, day 93.
  Weight (g)
Length | Day 1 (Baseline), Day 45, day 93.
  Length (cm)
Head Circumference | Day 1 (Baseline), Day 45, day 93.
  Head Circumference (cm)
Gastrointestinal tolerance | Day 7, day 24, day 45, day 52, day 73, day 93
  Numbers of Regurgitations, gassiness, rejections- Differences between groups measured by a 1-day record
Intestinal habits | Day 7, day 24, day 45, day 52, day 73, day 93
  Frequency of defecations and stools consistency- Differences between groups measured by 1-day record
Satiety | Day 7, day 24, day 45, day 52, day 73, day 93
  Food intake (amount), crying (time) and sleeping (time)-Differences between groups measured by 1-day record
Prebiotic effects | Day 1 (baseline), day 45
  Microbiome sequencing- Differences between groups measured in collected stools

CONTACTS AND LOCATIONS:
Overall Officials: David Gil, PhD, Principal Investigator — Hospital Virgen de la Arrixaca; Luis M Sánchez, PhD, Study Chair — Hero
Locations (4):
- Spain (4):
  - Institute Hero for Infant Nutrition, Alcantarilla, Murcia
  - Quantum Experimental, Murcia, Murcia
  - University of Murcia, Murcia, Murcia
  - Hospital Virgen de la Arrixaca, Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernal MJ, Periago MJ, Martinez R, Ortuno I, Sanchez-Solis M, Ros G, Romero F, Abellan P. Effects of infant cereals with different carbohydrate profiles on colonic function--randomised and double-blind clinical trial in infants aged between 6 and 12 months--pilot study. Eur J Pediatr. 2013 Nov;172(11):1535-42. doi: 10.1007/s00431-013-2079-3. Epub 2013 Jun 29. PMID 23812516
- [Result] Fardet A. New hypotheses for the health-protective mechanisms of whole-grain cereals: what is beyond fibre? Nutr Res Rev. 2010 Jun;23(1):65-134. doi: 10.1017/S0954422410000041. Epub 2010 Jun 22. PMID 20565994
- [Result] Stephen A, Alles M, de Graaf C, Fleith M, Hadjilucas E, Isaacs E, Maffeis C, Zeinstra G, Matthys C, Gil A. The role and requirements of digestible dietary carbohydrates in infants and toddlers. Eur J Clin Nutr. 2012 Jul;66(7):765-79. doi: 10.1038/ejcn.2012.27. Epub 2012 Apr 4. PMID 22473042
- [Result] Mennella JA, Trabulsi JC. Complementary foods and flavor experiences: setting the foundation. Ann Nutr Metab. 2012;60 Suppl 2(Suppl 2):40-50. doi: 10.1159/000335337. Epub 2012 Apr 27. PMID 22555188